CLINICAL TRIAL: NCT05193227
Title: A Randomized Phase 2 Trial of ST-01 (Sustained-release Lidocaine Polymer Solution for Injection) in Subjects Undergoing Pelvic Surgery
Brief Title: Sustained Release Lidocaine for the Treatment of Postoperative Pain
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Sustained Therapeutics Inc. (Industry)
Responsible Party: Principal Investigator, David Harriman, Assistant Professor, Department of Urologic Sciences, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H20-00317
Record Dates: First submitted 2021-12-08; First posted 2022-01-14 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Pain; Postsurgical Pain
Keywords: pelvic surgery; scrotal surgery; inguinal incision; circumcision; hemorrhoidectomy; fistulotomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (ST-01) (Experimental): Administration of ST-01 as single-dose into the cutaneous, subcutaneous and fascia region of the surgical site and/or as nerve block.
  Interventions: Drug: ST-01
- Control (Standard of Care) (Active Comparator): Administration of Control (Lidocaine Hydrochloride Injection USP Xylocaine® or Bupivacaine Hydrochloride Injection USP Marcaine®) as single-dose into the cutaneous, subcutaneous and fascia region of the surgical site and/or as nerve block.
  Interventions: Drug: Control (Lidocaine Hydrochloride Injection USP Xylocaine® or Bupivacaine Hydrochloride Injection USP Marcaine®)

INTERVENTIONS:
Drug: ST-01 — Administration of up to 8 mL ST-01 (70 mg/mL lidocaine)
  Arms: Treatment (ST-01)
Drug: Control (Lidocaine Hydrochloride Injection USP Xylocaine® or Bupivacaine Hydrochloride Injection USP Marcaine®) — Administration of up to 3 mg/kg bupivacaine hydrochloride injection (0.25%) or up to 4.5mg/kg lidocaine hydrochloride injection (0.5-1%)
  Arms: Control (Standard of Care)

SUMMARY:
In this study, the investigators are testing a new formulation of lidocaine for its suitability in managing postoperative pain after pelvic (circumcision, inguinal, scrotal), perineal (hemorrhoidectomy) or perianal (fistulotomy) incisions. The new formulation ST-01 is a sustained release lidocaine formulation and is expected to provide pain relief over multiple days. Currently, the drug lidocaine is not available as an injectable slow-release formulation.

DETAILED DESCRIPTION:
The purpose of this study is to find out if a new sustained release lidocaine polymer formulation can provide effective postoperative pain control after surgery and lower opioid consumption.

A single dose of this new formulation ST-01 is administered as peri-neural injection and incisional deposition. The procedure is very comparable to the current standard of care procedure, where lidocaine solution (Lidocaine HCl 1% USP) is administered. However, the polymer solution ST-01 stays in the area of injection longer by forming a soft implant and could provide longer pain control.

The investigators' primary objective is to evaluate the efficacy of an injection of ST-01 to reduce subject-reported postoperative pain after surgery compared to standard of care. Secondary objectives are to determine the safety, frequency and total intake of opioid analgesic medication and frequency and total intake of non-opioid analgesic medication.

The clinical study is conducted at the Vancouver Prostate Centre and St. Paul's Hospital. Potential participants will undergo a screening period and will then be enrolled and randomized to either receive treatment (ST-01) or Control (Standard of Care) after surgery. Up to 120 study subjects will be enrolled and monitored over 30 days after surgery. Subjects will report their postsurgical pain and analgesic medication taken.

The primary endpoint and other continuous secondary endpoints will be compared with independent two-sample t-test if normally distributed and Wilcoxon rank-sum test if not normally distributed.

ELIGIBILITY:
Inclusion Criteria:

* Any sex, aged ≥ 19 years
* Indication to undergo an operation with a planned pelvic incision
* Able and willing to provide informed consent
* Stated willingness to comply with all study procedures and availability for the duration of the study
* If sexually active, is willing to use adequate birth control methods to prevent pregnancy over the course of the study

Exclusion Criteria:

* History of chronic pain conditions associated with the use of opioids or steroids
* Known allergic reactions to any components of the investigational product
* Active infection involving the surgical site
* Any contraindication to local anesthesia with lidocaine (e.g., known hypersensitivity to anesthetics of the amide type, known hypokalemia, complete heart block, anticoagulants (ASA permitted) antiarrhythmic medication)
* Use of prohibited medications (quinidine, procainamide, disopyramide, lidocaine, mexiletine, flecainide, propafenone, amiodarone, dronedarone, ibutilide, dofetilide, sotalol, vernakalant)
* Has participated in another clinical trial within 3 months prior to the Screening Visit or is planning to participate in another clinical trial during this trial period
* Has any other surgical or medical condition that, in the judgment of the clinical Investigator might warrant exclusion or be contraindicated for safety reason

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2026-04-27 (Estimated); Study Completion 2026-05-27 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of an injection of ST-01 to reduce subject-reported postoperative pain after surgery compared to standard of care | 3 days
  The mean area under the curve (AUC) of the visual analogue scale (VAS) of pain intensity scores through day 3 (AUC0-3) for ST-01 compared with standard of care (SOC).

SECONDARY OUTCOMES:
To evaluate the safety of an injection of ST-01 | 30 days
  The incidence of treatment-emergent adverse events (TEAEs) and TEAEs related to the study treatment
To compare the intake of opioid analgesic medication by subjects after an injection of ST-01 or standard of care | 3 days
  The mean total postoperative opioid consumption through 3 days for ST-01 compared to SOC
To compare the intake of non-opioid analgesic medication by subjects after an injection of ST-01 or standard of care | 3 days
  The mean total postoperative non-opioid consumption through 3 days for ST-01 compared to SOC

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Boniface, PhD, Study Director — Sustained Therapeutics Inc.
Locations (2):
- Canada (2):
  - Vancouver Prostate Centre, Vancouver, British Columbia
  - St. Pauls Hospital, Vancouver, British Columbia